CLINICAL TRIAL: NCT00216710
Title: Evaluation of the Healthy Families Alaska Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: State of Alaska Department of Health and Social Services (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 99-0155; Contract Number 067727
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Child Abuse
Keywords: Child abuse; Neglect; Home visitation; Program evaluation
MeSH Terms: interventions — House Calls

ARMS (2):
- Home Visited Mothers (Experimental): Mothers randomized to the home visited group received AK State-funded home visiting services. Frequency of home visits was determined by home visiting staff based on mothers' needs. Mothers could receive home visiting services until their child turned 3 years old
  Interventions: Behavioral: Home Visiting
- Control Mothers (No Intervention): Mothers randomized to the control group did not receive home visiting services, but were offered referrals to other community-based services, as was usual protocol with home visiting agencies were operating at capacity.

INTERVENTIONS:
Behavioral: Home Visiting
  Arms: Home Visited Mothers

SUMMARY:
This study will assess the effectiveness of early home visitation by a professional in preventing child maltreatment, promoting healthy family functioning, and promoting child health and development.

The investigators will test the following hypotheses regarding the effectiveness of early paraprofessional home visiting for at-risk families

* Actual home visiting services adhere to HFAK standards.
* HFAK promotes healthy family functioning, promotes child health and development, and prevents child abuse and neglect.
* Adherence to HFAK process standards is positively associated with achievement of outcomes.

DETAILED DESCRIPTION:
Healthy Families Alaska (HFAK) is a well-established child abuse prevention program targeted to at-risk families. HFAK is based on the Healthy Families America initiative promoted by Prevent Child Abuse America. The State Department of Health and Social Services (DHSS) administers the HFAK program.

In 1998, the Alaska State Legislature requested a controlled study of HFAK to determine its effectiveness in preventing child maltreatment, promoting healthy family functioning, and promoting child health and development. DHSS awarded the Johns Hopkins University School of Medicine a contract to conduct the study from July 1999 through June 2004.

The study is a randomized trial of six HFAK sites throughout Alaska. It aims to compare services actually provided to HFAK standards, assess program success in achieving intended outcomes, and relate program impact to service delivery.

Families are enrolled over 21 months beginning in January 2000. Families are randomized to either the HFAk group or the control group. Baseline data on family attributes are collected from HFAK files and maternal interviews. HFAK service data are collected from the program's management information system, record reviews, surveys of staff, and staff focus groups. Outcome data are collected when the children were two years old through maternal interview, home-based observations, child developmental testing, review of medical records, and review of OCS child welfare records.

ELIGIBILITY:
Inclusion Criteria:

* Family resides in a community served by one of six HFAK programs participating in the study
* Family identified as at-risk by HFAK staff following the usual HFAK protocol

Exclusion Criteria:

* Family was previously enrolled in HFAK
* Mother unable to speak English well enough to complete study activities.
* Family unwilling to enroll in the HFAK program.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 1999-07; Primary Completion 2004-02-21 (Actual); Study Completion 2005-01-21 (Actual)

PRIMARY OUTCOMES:
Child Abuse and Neglect | From child's birth (baseline) to 24 months of age
  Substantiated and unsubstantiated reports of abuse; maternal self-report of harsh discipline
Child Development | 24 months
  Child cognitive, motor and psychosocial development

SECONDARY OUTCOMES:
Child Health | From child's birth (baseline) to 24 months of age
  Hospitalizations, ED use, injuries requiring medical care, adequate well child care, immunizations
Maternal Life Course | At time of study follow-up (child 24 months of age)
  Educational attainment, employment, social support, rapid repeat birth
Maternal Psychosocial Functioning | At time of study follow-up (child 24 months of age)
  Mental health, substance use, intimate partner violence
Parenting Knowledge | At time of study follow-up (child 24 months of age)
  Knowledge of child development; recognition of child delay
Parenting Attitudes | At time of study follow-up (child 24 months of age)
  Use of corporal punishment, infant caregiving, expectations of children, empathy towards child's needs
Parenting Behavior | At time of study follow-up (child 24 months of age)
  Observational measures of parent/child interaction and quality of the home environment, use of corporal punishment, use of nonviolent discipline

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Duggan, ScD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Anchorage, Alaska, United States